CLINICAL TRIAL: NCT02371759
Title: Efficacy and Safety of Intraoral Local Anesthesia by Lidocaine + Clonidine in Patients With Diabetes Mellitus Type 2
Brief Title: Lidocaine + Clonidine for Intraoral Anesthesia in Patients With Diabetes Mellitus Type 2
Acronym: LCIOADMT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Bozidar Brkovic, DDS, MSc, PhD, Professor, Professor, DDS, MSc, PhD, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UBelgrade 534/2; 175021 (Other Grant/Funding Number: Ministry of Education, Science and Technological Development)
Record Dates: First submitted 2015-02-04; First posted 2015-02-26 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus; Local Anesthesia
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Diabetics: L+C maxillary anesthesia (Experimental): Single dose intraoral local anesthesia with 2ml lidocaine (2%) + clonidine (15 mcg/ml) for maxillary infiltration anesthesia
  Interventions: Drug: L+C maxillary anesthesia
- Diabetics: L+C mandibular anesthesia (Experimental): Single dose intraoral local anesthesia with 2ml lidocaine (2%) + clonidine (15 mcg/ml) for mandibular block anesthesia
  Interventions: Drug: L+C mandibular anesthesia
- Diabetics: L+E maxillary anesthesia (Active Comparator): Single dose intraoral local anesthesia with 2ml lidocaine (2%)+ epinephrine (1:80.000) for maxillary infiltration anesthesia
  Interventions: Drug: L+E maxillary anesthesia
- Diabetics: L+E mandibular anesthesia (Active Comparator): Single dose intraoral local anesthesia with 2ml lidocaine (2%) + epinephrine (1:80.000) for mandibular block anesthesia
  Interventions: Drug: L+E mandibular anesthesia
- Healthy: L+C maxillary anesthesia (Experimental): Single dose intraoral local anesthesia with 2ml lidocaine (2%) + clonidine (15 mcg/ml) for maxillary infiltration anesthesia
  Interventions: Drug: L+C maxillary anesthesia
- Healthy: L+C mandibular anesthesia (Experimental): Single dose intraoral local anesthesia with 2ml lidocaine (2%) + clonidine (15 mcg/ml) for mandibular block anesthesia
  Interventions: Drug: L+C mandibular anesthesia
- Healthy: L+E maxillary anesthesia (Active Comparator): Single dose intraoral local anesthesia with 2ml lidocaine (2%)+ epinephrine (1:80.000) for maxillary infiltration anesthesia
  Interventions: Drug: L+E maxillary anesthesia
- Healthy: L+E mandibular anesthesia (Active Comparator): Single dose intraoral local anesthesia with 2ml lidocaine (2%) + epinephrine (1:80.000) for mandibular block anesthesia
  Interventions: Drug: L+E mandibular anesthesia

INTERVENTIONS:
Drug: L+C maxillary anesthesia — Maxillary anesthesia obtained by 2% lidocaine + clonidine (15 mcg/ml)
  Arms: Diabetics: L+C maxillary anesthesia; Healthy: L+C maxillary anesthesia
Drug: L+C mandibular anesthesia — Mandibular anesthesia obtained by 2% lidocaine + clonidine (15 mcg/ml)
  Arms: Diabetics: L+C mandibular anesthesia; Healthy: L+C mandibular anesthesia
Drug: L+E maxillary anesthesia — Maxillary anesthesia obtained by 2% lidocaine + epinephrine (1:80 000)
  Arms: Diabetics: L+E maxillary anesthesia; Healthy: L+E maxillary anesthesia
Drug: L+E mandibular anesthesia — Mandibular anesthesia obtained by 2% lidocaine + epinephrine (1:80 000)
  Arms: Diabetics: L+E mandibular anesthesia; Healthy: L+E mandibular anesthesia

SUMMARY:
The purpose of this study is to determine whether 2% lidocaine (L) + clonidine (C) (15 mcg/ml) as a vasoconstrictor achieves efficient (equal or better parameters of intraoral local anesthesia in comparison to 2% lidocaine + epinephrine (E) (1:80 000)) and safe (stable cardiovascular parameters - systolic, diastolic, mean blood pressure and heart rate) intraoral local anesthesia in patients with Diabetes mellitus type 2.

DETAILED DESCRIPTION:
Patients with diabetes mellitus type 2, represent a risk for performing regional anesthesia techniques due to microvascular (microangiopathy, neuropathy) and macrovascular (hypertension, coronary heart disease) complications. There is evidence that local anesthetic toxicity may be increased in diabetic setting due to underlying neuropathy; while interaction of diabetic blood vessels with vasoconstrictors may be of importance because of microangiopathic changes. Lately, regional anesthesia protocol in general surgery for patients with diabetes mellitus was released, proposing reduction of local anesthetic concentration and avoiding epinephrine as vasoconstrictor.

Oral cavity tissues in diabetes mellitus also suffer from neuropathy (burning, paresthesia, teeth loss, temporomandibular dysfunction, xerostomia) and microangiopathy (periodontal disease, salivary gland dysfunction). Most widely used vasoconstrictor for intraoral local anesthesia, epinephrine, is an alpha- and beta- adrenergic agonist. Because of its beta-adrenergic effects, epinephrine could adversely affect cardiovascular function, especially in risk patients. There are data suggesting that intraoral local anesthesia obtained with 2% lidocaine with clonidine, selective alpha 2-adrenoceptor agonist as a vasoconstrictor, is characterized with significantly more stable cardiovascular parameters and similar parameters of local anesthesia with respect to lidocaine with epinephrine in healthy and hypertensive patients.

With regard to aforementioned, the aim of this randomized double-blind controlled clinical trial is to evaluate and compare efficacy and safety of intraoral local anesthesia obtained with 2% lidocaine (L) + clonidine (15 mcg/ml) (C) or 2% L + epinephrine (1:80 000) (E), comparing healthy and diabetes mellitus type 2 patients. Prior to tooth extraction, random allocation to one of four groups (L+C maxillary infiltration, L+C mandibular block, L+E maxillary infiltration and L+E mandibular block) is performed for diabetic (30 per group) and healthy (30 per group) patients. Parameters of local anesthesia (onset, duration, intensity, width of anesthetic field for maxillary infiltration), cardiovascular parameters (systolic, diastolic, mean arterial pressure; heart rate and electrocardiographic changes), quality of postoperative analgesia (assessed by Visual Analogue Scale, Numerical Rating Scale and number of consumed analgesics) and postoperative complications (infection, bleeding, paresthesia, delayed wound healing) are evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants: ASA I
* Diabetic type 2 participants: ASA III (HbA1c level < 9%)
* Required a single-root teeth indicated for non-complicated extraction
* Dental diagnosis of periodontal disease, tooth fracture, chronic periapical lesion and root infection
* Subjects give informed written consent

Exclusion Criteria:

* Pregnancy and lactation
* Allergy to used drugs and food
* Hepatic and/or renal failure
* ASA IV patients
* Tobacco smokers
* History of alcoholism and/or drug abuse and addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragica DM Stojic, DDS, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade; Bozidar M Brkovic, DDS, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade; Marija S Milic, DDS, Principal Investigator — School of Dental Medicine, University of Belgrade
Locations (1):
- School of Dental Medicine, University of Belgrade, Belgrade, Serbia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between june 2013 and december 2015 among the patients of Clinic of Oral Surgery, Faculty of Dental Medicine, University of Belgrade
Period: Overall Study
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Started | 32 | 31 | 33 | 31 | 27 | 26 | 25 | 28
Completed | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Not Completed | 3 | 1 | 1 | 0 | 3 | 1 | 0 | 4
Not completed — Protocol Violation | 3 | 1 | 1 | 0 | 3 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia | Total
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24 | 220
Age, Categorical [Count of Participants; unit: Participants] — Age between 18 and 65 years
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24 | 220
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 21 | 14 | 9 | 15 | 15 | 14 | 126
  Male | 7 | 14 | 11 | 17 | 15 | 10 | 10 | 10 | 94
Region of Enrollment [Number; unit: participants]
  Serbia | 32 | 31 | 33 | 31 | 24 | 25 | 25 | 24 | 220
Body Mass [Mean (Standard Deviation); unit: kilograms] | 78.72 (11.19) | 75.03 (11.53) | 85.84 (14.76) | 79.45 (17.34) | 79.50 (15.22) | 74.59 (9.64) | 71.01 (12.08) | 71.59 (7.81) | 76.90 (8.42)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: milimoles per liter] — Available only for diabetic participants
  milimoles per liter | 8.12 (3.01) | 7.55 (2.53) | 9.66 (4.02) | 8.35 (2.49) | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.83 (4.59) | 9.57 (5.51) | 9.77 (7.62) | 9.27 (6.09) | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants
Glycosilated Hemoglobin [Mean (Standard Deviation); unit: percents] | 7.42 (1.25) | 7.55 (2.53) | 7.63 (1.72) | 7.97 (1.50) | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants | NA (NA) — Available only for diabetic participants
Number of participants with modified diet [Count of Participants; unit: Participants] | 22 | 30 | 31 | 30 | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Total not calculated because data are not available (NA) in one or more arms.
Number of participants on OHA therapy [Count of Participants; unit: Participants] | 28 | 29 | 30 | 30 | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Total not calculated because data are not available (NA) in one or more arms.
Number of participants on insulin therapy [Count of Participants; unit: Participants] | 2 | 4 | 8 | 4 | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Total not calculated because data are not available (NA) in one or more arms.
Hypertension [Count of Participants; unit: Participants] | 16 | 26 | 19 | 17 | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Total not calculated because data are not available (NA) in one or more arms.
Coronary Artery Disease [Count of Participants; unit: Participants] | 12 | 14 | 14 | 13 | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Total not calculated because data are not available (NA) in one or more arms.
Peripheral Neuropathy [Count of Participants; unit: Participants] | 9 | 12 | 12 | 10 | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Total not calculated because data are not available (NA) in one or more arms.
Intraoral Neuropathy [Count of Participants; unit: Participants] | 14 | 16 | 17 | 18 | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Available only for diabetic participants | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Duration of Intraoral Local Anesthesia
Description: Time until cessation in soft tissue numbness
Time Frame: Up to 6 hours after local anesthesia injection
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
minutes | 132.48 (91.86) | 173.27 (70.44) | 182.09 (57.86) | 195.35 (68.99) | 108.82 (27.76) | 155.59 (60.75) | 114.74 (39.72) | 172.91 (68.93)
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; In order to detect 20% difference in intraoral anesthesia duration between healthy and diabetic participants, with 80 % statistical power at a two-tailed significance level of 0.05 using Mann Whitney U test, it was calculated that at least 24 participants must be included in each group; Test type: Non-Inferiority or Equivalence — In order to detect 20% difference in intraoral anesthesia duration between healthy and diabetic participants, with 80 % statistical power at a two-tailed significance level of 0.05 using Mann Whitney U test, it was calculated that at least 24 participants must be included in each group; p < 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Intensity of Intraoral Local Anesthesia
Description: Number of participants who reported values > 0 after pin-prick testing, using Visual Analogue Scale (VAS) and Numerical Rating Scale (NRS). VAS is represented by line 100 mm long, with one end marked with 0 and words "no pain" , while the other end is marked with 100 and words "the worst pain imanginable". VRS scale is represented by line 100 mm long, marked with numbers from 0 to 10, where 0 corresponds to "no pain", and 10 corresponds to "the worst pain imaginable". For both scales, higher scores represent worse outcomes.
Time Frame: Up to 10 minutes after local anesthesia injection
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Participants | 2 | 2 | 1 | 8 | 2 | 1 | 4 | 6
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Chi-squared

3. Primary Outcome: Baseline Systolic Blood Pressure
Time Frame: Baseline, 0 minutes
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 135.2759 (16.69665611) | 137.7333 (18.43335308) | 134.8125 (18.66934265) | 134.4667 (17.69119729) | 124.0455 (11.07325079) | 128.1818 (15.49388931) | 125 (11.11918898) | 126.5909 (18.82322642)

4. Primary Outcome: Systolic Blood Pressure at 10 Minutes
Description: Systolic blood pressure values 5 minutes after local anesthesia injection
Time Frame: 10th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 130.3793 (18.81377496) | 136.8333 (14.27098173) | 137.4375 (19.73033934) | 132.6 (20.45858857) | 120.8182 (13.58092627) | 122.5909 (14.59503859) | 125.8261 (13.75979708) | 125,4091 (12.71541656)

5. Primary Outcome: Systolic Blood Pressure at 15 Minutes
Description: Systolic blood pressure values 10 minutes after local anesthesia injection
Time Frame: 15th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 133.5862 (13.51590925) | 133.4667 (14.12684735) | 137.4688 (19.28058421) | 132.0667 (17.89580957) | 114.4545 (11.89128241) | 116.9091 (12.78730431) | 123.8696 (13.61250878) | 127.1818 (18.58733917)

6. Primary Outcome: Systolic Blood Pressure at 20 Minutes
Description: Systolic blood pressure values 15 minutes after local anesthesia injection
Time Frame: 20th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 130.2414 (14.98011819) | 131.3333 (14.73755076) | 132.4063 (17.69428443) | 133.2333 (18.46560212) | 108.8182 (9.529630256) | 120.8636 (12.995587) | 123.8696 (12.15918788) | 124.6818 (19.56767588)

7. Primary Outcome: Systolic Blood Pressure at 35 Minutes
Description: Systolic blood pressure values 30 minutes after local anesthesia injection
Time Frame: 35th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 127.2759 (12.91979807) | 130.3 (13.12841089) | 132.5625 (17.0330561) | 132.7 (16.38723706) | 116.3636 (7.364945637) | 120.1364 (14.54809906) | 120.6522 (10.01185069) | 126.4545 (17.25916533)

8. Primary Outcome: Baseline Diastolic Blood Pressure
Time Frame: baseline, 0 minutes
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 74.1379 (11.37894088) | 81.7667 (9.722648048) | 75.25 (12.09372004) | 79.2 (15.61345574) | 73.1364 (9.627814144) | 80.9545 (11.23547644) | 76.3913 (5.694807287) | 75.0909 (12.72758194)

9. Primary Outcome: Diastolic Blood Pressure at 10 Minutes
Description: Diastolic blood pressure values 5 minutes after local anesthesia injection
Time Frame: 10th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 74.0345 (8.398480979) | 75.3667 (12.09830424) | 75.6875 (14.74829132) | 79.1 (15.23497999) | 69.7273 (10.49798991) | 75.0909 (6.560408603) | 75.8261 (7.010720193) | 73.8636 (10.14793178)

10. Primary Outcome: Diastolic Blood Pressure at 15 Minutes
Description: Diastolic blood pressure values 10 minutes after local anesthesia injection
Time Frame: 15th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 72.6897 (6.876998142) | 74.8 (9.672154605) | 74.8125 (13.17729597) | 80.0333 (13.86217876) | 69.3636 (9.800609576) | 72.5 (7.163066648) | 79 (15.45374329) | 74.1818 (11.57434093)

11. Primary Outcome: Diastolic Blood Pressure at 20 Minutes
Description: Diastolic blood pressure values 15 minutes after local anesthesia injection
Time Frame: 20th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 71.6897 (7.865400945) | 74.1667 (9.013718791) | 74.1563 (11.65390527) | 80.8333 (13.56465997) | 69.4545 (6.200823853) | 75.9545 (8.566141948) | 77 (9.060403362) | 76.0455 (14.81144111)

12. Primary Outcome: Diastolic Blood Pressure at 35 Minutes
Description: Diastolic blood pressure values 30 minutes after local anesthesia injection
Time Frame: 35th minute
Measure: Mean (Standard Deviation); unit: milimeters of Hg
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters of Hg | 70.1379 (8.140393716) | 74.3667 (10.37021597) | 73.2813 (12.59091935) | 75.9 (12.29859279) | 69.1364 (7.146730552) | 77.0455 (7.587441207) | 77.6087 (7.19051857) | 74.7273 (8.446931357)

13. Primary Outcome: Baseline Values of Heart Rate
Time Frame: baseline, 0 minutes
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
beats per minute | 75.0345 (10.80172856) | 80.7727 (6.682366571) | 78.3438 (10.20312847) | 84.2581 (13.16806172) | 76.4545 (14.44769638) | 73.0333 (8.695547948) | 76.2174 (14.04031463) | 76.3636 (9.756782523)

14. Primary Outcome: Heart Rate at 10 Minutes
Description: Heart rate 5 minutes after local anesthesia injection, 10 minutes after baseline measurement
Time Frame: 10th minute
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
beats per minute | 75.3448 (11.45262248) | 81.7727 (5.72311305) | 83.3125 (10.35012077) | 88.5806 (12.72209153) | 74.0455 (15.06012481) | 73.0667 (7.671417688) | 83.913 (14.36811358) | 83.6818 (13.23554508)

15. Primary Outcome: Heart Rate at 15 Minutes
Description: Heart rate 10 minutes after local anesthesia injection, 15 minutes after baseline measurement
Time Frame: 15th minute
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
beats per minute | 73.0345 (10.10828076) | 77.4545 (6.790883003) | 83.4688 (10.92196477) | 86.8387 (12.41261932) | 74.5 (12.91271061) | 73.4333 (4.896327805) | 81.6957 (14.48974013) | 83.5909 (11.09121957)

16. Primary Outcome: Heart Rate at 20 Minutes
Description: Heart rate 15 minutes after local anesthesia injection, 20 minutes after baseline measurement
Time Frame: 20th minute
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
beats per minute | 72.2414 (9.697772839) | 80.2273 (7.276477612) | 81.3125 (11.56032565) | 86.1935 (12.04552297) | 73.6818 (12.32645766) | 71.8667 (5.281881142) | 79.8435 (13.46448997) | 82 (11.84824681)

17. Primary Outcome: Ceart Rate at 35 Minutes
Description: Heart rate 30 minutes after local anesthesia injection, 35 minutes after baseline measurement
Time Frame: 35th minute
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
beats per minute | 72.1034 (9.236359934) | 80.8182 (6.095127129) | 80.0938 (11.04348991) | 85.3871 (11.87062879) | 71.3636 (12.53393662) | 73.4333 (7.762157062) | 77 (13.78017709) | 78.2273 (12.75382974)

18. Primary Outcome: Baseline Electrocardiogram
Time Frame: baseline, 0 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Chi-squared

19. Primary Outcome: Electrocardiogram at 10 Minutes
Description: ECG 5 minutes after local anesthesia injection, 10 minutes after baseline measurement
Time Frame: 10th minute
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Chi-squared

20. Primary Outcome: Electrocardiogram at 15 Minutes
Description: ECG 10 minutes after local anesthesia injection, 15 minutes after baseline measurement
Time Frame: 15th minute
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Chi-squared

21. Primary Outcome: Electrocardiogram at 20 Minutes
Description: ECG 15 minutes after local anesthesia injection, 20 minutes after baseline measurement
Time Frame: 20th minute
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Chi-squared

22. Secondary Outcome: Onset of Intraoral Local Anesthesia
Description: Evaluated by pin-prick after subjective feeling of soft tissue numbness appeared after local anesthesia injection
Time Frame: Up to 10 minutes, until subjective feeling of soft tissue numbnes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 25
minutes | 1.76 (0.87) | 5.27 (2.12) | 2.16 (1.08) | 5.45 (2.64) | 2.77 (1.11) | 4.59 (2.58) | 2.83 (0.83) | 6.36 (2.3)
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Width of Anesthetic Field After Maxillary Infiltration Anesthesia
Description: Soft tissue numbness area determined by pin-prick test after maxillary infiltration anesthesia. Not tested for mandibular ablock anesthesia.
Time Frame: Up to 10 minutes after injection of local anesthesia
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
milimeters | 27.07 (1.06) | NA (NA) — Measured only after infiltration technique | 35.19 (1.67) | NA (NA) — Measured only after infiltration technique | 23.81 (1.07) | NA (NA) — Measured only after infiltration technique | 24.52 (0.95) | NA (NA) — Measured only after infiltration technique
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+E Maxillary Anesthesia; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney)

24. Secondary Outcome: Postoperative Analgesia
Description: Number of participants who experienced postoperative pain, VAS, NRS
Time Frame: up to 24 hours after tooth extraction
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Participants | 11 | 15 | 13 | 14 | 5 | 14 | 10 | 12
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Chi-squared

25. Secondary Outcome: Local Postoperative Complications
Description: Postoperative paresthesia by clinical examination
Time Frame: 24 hours, 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Number analyzed (Participants) | 29 | 30 | 32 | 31 | 24 | 25 | 25 | 24
Participants | 1 | 1 | 6 | 4 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Diabetics: L+C Maxillary Anesthesia vs Diabetics: L+C Mandibular Anesthesia vs Diabetics: L+E Maxillary Anesthesia vs Diabetics: L+E Mandibular Anesthesia vs Healthy: L+C Maxillary Anesthesia vs Healthy: L+C Mandibular Anesthesia vs Healthy: L+E Maxillary Anesthesia vs Healthy: L+E Mandibular Anesthesia; Test type: Superiority or Other; p < 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Diabetics: L+C Maxillary Anesthesia | Diabetics: L+C Mandibular Anesthesia | Diabetics: L+E Maxillary Anesthesia | Diabetics: L+E Mandibular Anesthesia | Healthy: L+C Maxillary Anesthesia | Healthy: L+C Mandibular Anesthesia | Healthy: L+E Maxillary Anesthesia | Healthy: L+E Mandibular Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/32 | 0/31 | 0/24 | 0/25 | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/32 | 0/31 | 0/24 | 0/25 | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes